CLINICAL TRIAL: NCT04223934
Title: ARTERY Outcomes: Tailored Drug Titration Through Artificial Intelligence - an Interventional Study
Brief Title: Tailored Drug Titration Using Artificial Intelligence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optima Integrated Health (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O4BP-001
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized, intervention versus control.
Who Masked: Participant
Masking Description: Patient blinded to assignment [intervention versus control].
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optima4BP (Experimental): Treating physicians receive periodic (every 5-8 weeks) medication treatment recommendations intended to optimize the current patient treatment.
  The recommendations are generated based on periodic remote data collected from the patient and from the Electronic Health Record. The analysis of the data allows assessment of the patient's response to current treatment and need for a treatment optimization. If a treatment optimization is needed, one is generated and sent to the treating physician for consideration.
  Interventions: Other: optima4BP
- Standard of Care (SOC) (No Intervention): The treating physician follows usual care practices.

INTERVENTIONS:
Other: optima4BP — optima4BP establishes a "no gaps" computational framework in determining the most effective treatment change that can optimize a patient's HTN management towards BP Target. All possible drug combination options available through the 16 anti-HTN drug classes and subclasses are quantitatively evaluated in the context of 5 actions: add a drug, remove a drug, replace a drug, increase a drug dose, and decrease a drug dose. The pharmacological intervention efficacy ranking is computed and the highest ranked treatment recommendation is selected for consideration by the treating physician.
  Arms: optima4BP

SUMMARY:
The purpose of the ARTERY Outcomes study is to compare optima-for-blood pressure (optima4BP), a clinical decision support system for hypertension (HTN) treatment optimization to standard of care in patients with essential HTN.

DETAILED DESCRIPTION:
Nearly 34 million Americans have their blood pressure (BP) uncontrolled. Hypertension (HTN) claims 1000 deaths every day. Despite medication and life-style management, the cost of HTN associated hospitalizations had escalated to $113 billion in 2016, or 15% of all hospital costs, with >135 million Emergency Department (ED) visits.

Uncontrolled HTN for even a few weeks is associated with increased risk for acute cardiovascular (CVD) events [stroke, heart failure (HF), myocardial infarction (MI)] and death. Medication treatment optimization to BP goal reduces the incidence of stroke by 35-40%, HF by up to 64%, and MI by 15-25%.

optima-for-blood pressure [optima4BP] transforms the episodic and reactive nature of uncontrolled HTN pharmacological treatment management into a process that is continuous, proactive, and personalized. The innovation simulates the established clinical reasoning treatment decision process undertaken during a patient's visit.

ELIGIBILITY:
Inclusion Criteria:

* Two or more blood pressure (BP) readings of ≥ 140/90 mmHg during UCSF primary care or cardiology office visits within the last 12 months
* Therapy with medications from at least 1 anti-HTN pharmacological agents at the time of the last office visit
* At least minimally "tech-savvy" defined as Ownership of a compatible smartphone and Ability to access the internet
* Active Electronic Health Record MyChart account

Exclusion Criteria:

* Home anti-HTN medication therapy doesn't match the electronic health record medication list
* Anti-HTN medication therapy changed within 30 days prior to enrollment
* Inability to operate a BP cuff
* Incompatible smartphone device (Galaxy S5 Android 5.0)
* Less than minimally "tech-savvy" defined as Inability to use the Internet
* Non-compliance with medical follow-up (>3 "no shows" in the previous 12 months)
* Planned coronary revascularization in the next 12 months
* Myocardial infarction, coronary revascularization, stroke, cardiac or aortic surgery in the previous 90 days
* GFR < 30 (CKD stage IV/ V)
* Treating physician rules out the patient due to superseding health management concerns
* Treating physician rules out the patient due to other concerns

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Reduction in systolic BP [SBP] (mmHg) measured remotely [Time frame: 0 - 6 months] | 6 months
  optima4BP leads ≥4mmHg of SBP reduction compared to Standard of Care

SECONDARY OUTCOMES:
Incidence of Adverse Events [Time Frame: full 12 months] | 6 months and 12 months
  Frequency and severity of adverse events (AEs) between baseline and the end of the study.
Sustained remote SBP Target during observational period [Time Frame: 6 - 12 months (end of study)] | 6 months
  Without optima4BP intervention, the O4BP arm will maintain a ≥4mmHg remote systolic blood pressure (SBP) reduction compared to the SOC arm

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Voskerician, PhD, Study Director — Optima Integrated Health; Liviu Klein, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be made available to other researchers.